CLINICAL TRIAL: NCT01037725
Title: A Phase-1, Single Center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics (Including Food Effect) of Ascending Oral Doses of AZD5847 in Healthy Male Subjects and Female Subjects of Non-childbearing Potential
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics (PK) (Including Food Effect) of Oral Doses of AZD5847 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D3430C00001
Record Dates: First submitted 2009-12-20; First posted 2009-12-23 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Healthy volunteer; first time in human; food effect
MeSH Terms: interventions — posizolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD5847 oral suspension (Experimental): Active
  Interventions: Drug: AZD5847
- Placebo to AZD5847 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo to AZD5847

INTERVENTIONS:
Drug: AZD5847 — Part A - Oral doses given to approximately 6 cohorts of 8 subjects (6 on active and 2 on placebo) on Day 1.
  Part B - Oral doses of AZD5847 given to 1 cohort of 8 subjects on Days 1 and 8 in either a fasted state or with a high fat meal
  Arms: AZD5847 oral suspension
Drug: Placebo to AZD5847 — In Part A - Single oral doses of AZD5847placebo given to approximately 6 cohorts of 8 subjects each (6 on active and 2 on placebo) on Day 1
  Arms: Placebo to AZD5847

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of AZD5847 after receiving oral doses on a single day (Part A) or after receiving a single oral dose in two periods (Part B). For volunteers in Part B, the effect of food on the PK of AZD5847 will also be studied. Another purpose is to evaluate the pharmacokinetics (PK) of AZD5847 and its metabolites in blood and urine.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures
* Clinically normal physical findings and laboratory values as judged by the investigator with normal ECG.
* Healthy male and female volunteers. Females must be of non childbearing potential

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the investigator, within 4 weeks of the first administration of the Investigational Product
* History of any disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-12; Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD5847 administered orally will be assessed by incidence and severity of AE's, abnormalities in vital sign assessments, ECG's, telemetry, clinical laboratory assessments, physical exams and withdrawals | Safety assessments are taken prior to and after drug administration. Volunteers will be monitored througout the study for adverse events.

SECONDARY OUTCOMES:
To characterize the pharmacokinetics of AZD5847 in blood and urine following oral doses. | Samples taken during the residential period at defined timepoints pre-dose and post-dose.
To assess the effect of food on the pharmacokinetics of AZD5847 following oral administration of AZD5847 | Samples taken during the residential period at defined timepoints pre-dose and post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Patricia A Meier, MSc, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States